CLINICAL TRIAL: NCT03811067
Title: Transversus Abdominis Plane Block Versus Rectus Sheath Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane Block Versus Rectus Sheath Block After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hadi Ufuk Yörükoğlu, Principal investigator, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KAEK 2017/348
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Transversus abdominis plane block; Rectus sheath block; Cesarean delivery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- TAP group (Active Comparator): Transversus abdominis plane block administered group
  Interventions: Procedure: Transversus abdominis plane block
- RS group (Active Comparator): Rectus sheath block administered group
  Interventions: Procedure: Rectus sheath block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — Transversus abdominis plane block will be performed bilaterally after the surgery.
  Arms: TAP group
Procedure: Rectus sheath block — Rectus sheath block will be performed bilaterally after the surgery.
  Arms: RS group

SUMMARY:
Importance of effective postoperative pain management is well known. The undesired effects of pain can be prevented with multimodal analgesia for the patient. Overall, for cesarean delivery, interaction between the mother and her newborn baby can be provided earlier. Many regional anesthesia techniques can be prefferred after cesarean delivery. Aim of the study is to compare the postoperative analgesia effects of transversus abdominis plane block and rectus sheath block after elective cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II patients Patients undergo elective cesarean delivery Gestation period between 37-40 weeks

Exclusion Criteria:

obesity (body mass index >35 kg/m2) infection of the skin at the site of needle puncture area patients with known allergies to any of the study drugs coagulopathy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative 24th hour.
  Morphine consumption (mg) of patients with patient controlled device
NRS score | Postoperative 24th hour
  Numerating rating scale of patients

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Ufuk MD Yörükoğlu, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No